CLINICAL TRIAL: NCT03510390
Title: Metformin in Head and Neck Squamous Cell Carcinoma: A Window of Opportunity Study to Assess the Effect on Tissue Oxygenation
Brief Title: Metformin in Head and Neck Squamous Cell Carcinoma: Effect on Tissue Oxygenation
Acronym: HEAD-MET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: University of Bern (Other); Werner und Hedy Berger-Janser - Stiftung (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 3598
Record Dates: First submitted 2018-04-20; First posted 2018-04-27 (Actual); Last update posted 2021-11-18 (Actual); Status verified 2021-11

CONDITIONS: Head and Neck Cancer; Oral Cavity Squamous Cell Carcinoma
Keywords: head and neck cancer; tissue hypoxia; metformin
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Metformin

STUDY DESIGN:
Intervention Model Description: Window-of-opportunity
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Metformin (Experimental): Participants will be orally administered 850 mg of metformin twice daily between the therapeutic decision of the tumor board and the surgical resection of the tumor. The duration of the treatment is 9-14 days
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — 850 mg, oral, twice daily, 9-14 days

SUMMARY:
The study evaluates the effects of the drug Metformin on the oxygen content in cancer tissue. Low oxygen concentration in cancer tissue accelerates cancer growth. Moreover, the response to radiation therapy is worse when tissue oxygen is low, because radiation therapy depends on oxygen to unfold therapeutic effects. Metformin has been used to treat type II diabetes for over 50 years and features additional properties that could slow down cancer growth. One of these properties is the improved oxygen concentration in cancer tissue. This effect has been proven for various cancers.

This study was planned to verify this effect in head and neck cancer. Patients who suffer from cancer of the mouth and are planned for surgical removal of the cancer will be given Metformin for 9 to 14 days. The tissue removed in the subsequent surgery will be compared to a tissue sample that had been taken from the same patient prior to Metformin intake. To evaluate the oxygen content in the tissue samples, the expression of genes that react to oxygen levels will be measured and compared between the samples taken before and after treatment with Metformin.

A secondary aim is to evaluate whether changes in the oxygen content within the tumor can be visualized by means of magnetic resonance imaging (MRI). Therefore, participants undergo an MRI scan, before and after Treatment with Metformin. The changes in the MRI will be correlated to the changes measured in gene expression.

DETAILED DESCRIPTION:
The main objective of this trial is to prove the hypothesis that Metformin reduces tissue hypoxia in oral cavity squamous cell carcinoma after a course of treatment of 9-14 days.

The primary endpoint of the trial is the change in hypoxia-regulated gene expression upon Treatment with Metformin. Secondary endpoint are changes in MRI imaging correlating with the changes in gene expression.

Study design: This is a single-arm, open-label interventional window of opportunity study for proof of principle. Oral cavity squamous cell carcinoma is primarily treated by surgical tumor resection. This offers the possibility to study the effect of metformin on the tumor tissue.

Baseline tissue from potential participants before the intervention will be acquired by biopsy during diagnostic panendoscopy. Provided surgery is recommended by tumor board decision, participants will be orally administered 850 mg of metformin twice daily between the therapeutic decision of the tumor board and the surgical resection of the tumor. The duration of the treatment is 9-14 days, depending on the date of the planned surgery. The resected tumor tissue as well as the biopsy taken prior to metformin treatment will be subjected to massive parallel sequencing and immunohistochemistry.

To assess whether changes in hypoxia regulated gene expression can be correlated to changes in MRI scans, each participants will undergo a MRI scan before metformin treatment and a second MRI scan within 48 hours prior to the surgical resection of the tumor.

ELIGIBILITY:
Inclusion Criteria:

* Patients with biopsy-proven oral cavity squamous cell carcinoma, planned for tumor resection upon institutional tumor board decision.
* Tumor tissue (biopsy) prior to metformin administration available for genetic testing
* Age ≥ 18 years of age.
* First diagnosis, no prior treatment.
* All subjects must be able to comprehend and sign a written informed consent document.
* Informed consent as documented by signature

Exclusion Criteria:

* Pregnancy or lactation.
* Distant metastasis.
* Hypersensitivity to metformin or any of its components.
* Metformin treatment for any reason during the preceding 3 months.
* Diabetic patients regardless of treatment.
* Patients planned for imaging using iodinated contrast dye within 16 days prior to surgery.
* Any concomitant drug contraindicated for use with metformin according to the approved product information.
* Plasma alanine aminotransferase > 50 IU/dL.
* Plasma aspartate aminotransferase > 50 IU/dL.
* Estimated glomerular filtration rate (eGFR) <60 ml/min/1.73m2.
* Plasma alkaline phosphatase greater than 190 IU/dL.
* History of lactic or any other metabolic acidosis.
* History of diseases potentially causing tissue hypoxia and/or increased risk of lactic acidosis:
* Congestive heart failure.
* Myocardial ischemia within the last 6 months
* Sepsis or severe infection.
* History of lung disease currently requiring any pharmacologic or supplemental oxygen treatment.
* History of hepatic dysfunction or hepatic disease.
* Chronic alcoholism which poses a risk for acute alcohol intoxication at the discretion of the treating physician.
* Scheduled definitive surgical resection less than 10 days from enrollment.
* Any other serious underlying medical, psychiatric, psychological, familial or geographical condition, which in the judgment of the investigator may interfere with the planned staging, treatment, affect patient compliance or place the patient at high risk from treatment-related complication
* Known or suspected non-compliance.
* Participation in another study with investigational drug within the 30 days preceding and during the present study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2018-06-13 (Actual); Primary Completion 2021-09-15 (Actual); Study Completion 2021-11-15 (Actual)

PRIMARY OUTCOMES:
Metformin dependent changes in gene expression | Baseline and two weeks
  Metformin induced changes in gene expression between samples taken before and after the intervention, analyzed by RNAseq, with special attention to hypoxia responsive genes:
  * Hypoxia inducible factor 1 (HIF1) and co-transcription factors (ARNT, COPS5, HIF1A, HIFAN, HIF3a, HNF4A, NCOA1, PER1)
  * HIF interactors (APEX1, EGLN1, EGLN2, NFKB1, P4HA1, P4HB, TP53)
  * Markers of Angiogenesis (ADROA2B, ANGPTL4, ANXA2, BTG1, EGR1, EDN1, EPO, F3, GPI, HMOX1, JMJD6, LOX, MMP9, PGF, PLAU, SERPINE1, VEGFA)
  Additionally, metformin induced changes in HIF1A, Ki67, cleaved caspase 3, CAIX, p-mTOR and p-AKT will be assessed by immunohistochemistry

SECONDARY OUTCOMES:
Hypoxia dependent changes in MRI | baseline and two weeks
  Diffusion-weighted MRI and blood oxygen level dependent imaging (BOLD) will be obtained before and after the Intervention and compared. Alterations will be correlated to changes in gene Expression.

CONTACTS AND LOCATIONS:
Overall Officials: Olgun Elicin, MD, Principal Investigator — University Hospital Inselspital, Bern, Switzerland; Simon Mueller, MD, Principal Investigator — University Hospital Inselspital, Bern, Switzerland
Locations (1):
- Inselspital, Bern University Hospital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided